CLINICAL TRIAL: NCT01624090
Title: Phase II Evaluation of Mithramycin, an Inhibitor of Cancer Stem Cell Signaling, in Patients With Malignancies Involving Lungs, Esophagus, Pleura, or Mediastinum
Brief Title: Mithramycin for Lung, Esophagus, and Other Chest Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Schrump, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120151; 12-C-0151
Record Dates: First submitted 2012-06-16; First posted 2012-06-20 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer; Esophageal Cancer; Mesothelioma; Gastrointestinal Neoplasms; Breast Cancer
Keywords: Cancer Stem Cell; Thoracic Malignancies; Mithramycin Treatment; Lung Tumors; Metastatic Lung Tumors
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Mesothelioma; Gastrointestinal Neoplasms; Breast Neoplasms | interventions — Plicamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/mithramycin (Experimental): Single agent intravenous (IV) mithramycin
  Interventions: Drug: Mithramycin

INTERVENTIONS:
Drug: Mithramycin — 30 mcg/kg intravenous (IV) over 6 hours once daily for 7 days, to be repeated every 21 days (one cycle) until disease progression or unacceptable toxicity
  Other Names: Mithracin

SUMMARY:
Background:

- Mithramycin is a drug that was first tested as a cancer therapy in the 1960s. It acted against some forms of cancer, but was never accepted as a treatment. Research suggests that it may be useful against some cancers of the chest, such as lung and esophageal cancer or mesothelioma. Researchers want to see if mithramycin can be used to treat these types of cancer.

Objectives:

- To see if mithramycin is safe and effective against different chest cancers.

Eligibility:

- Individuals at least 18 years of age who have lung, esophagus, pleura, or mediastinum cancers.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and tumor tissue samples will be used to monitor the cancer before treatment.
* Participants will receive mithramycin every day for 7 days, followed by 7 days without treatment. Each 14-day round of treatment is called a cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take the drug for as long as the side effects are not severe and the tumor responds to treatment.

DETAILED DESCRIPTION:
Background:

Increasing evidence indicates that activation of stem cell gene expression is a common mechanism by which environmental carcinogens mediate initiation and progression of thoracic malignancies. Similar mechanisms appear to contribute to extra-thoracic malignancies that metastasize to the chest. Utilization of pharmacologic agents, which target gene regulatory networks mediating stemness may be novel strategies for treatment of these neoplasms. Recent studies performed in the Thoracic Epigenetics Laboratory, Thoracic and Oncology Surgery Branch (TOSB)/National Cancer Institute (NCI), demonstrate that under exposure conditions potentially achievable in clinical settings, mithramycin diminishes stem cell gene expression and markedly inhibits growth of lung and esophageal cancer and malignant pleural mesothelioma (MPM) cells in vitro and in vivo. These finding add to other recent preclinical studies demonstrating impressive anti-tumor activity of mithramycin in epithelial malignancies and sarcomas that frequently metastasize to the thorax.

Primary Objective:

-To assess clinical response rates of mithramycin administered as 6 hour intravenous infusions in patients with malignancies involving lungs, esophagus, pleura, or mediastinum.

Eligibility:

* Patients with measurable inoperable, histologically confirmed primary lung and esophageal carcinomas, thymic neoplasms, germ cell tumors, malignant pleural mesotheliomas or chest wall sarcomas, as well as patients with gastric, colorectal or renal cancers and sarcomas metastatic to the thorax are eligible.
* Patients with germline single nucleotide polymorphisms (SNPs) in adenosine 5-triphosphate binding cassette subfamily B member 4 (ABCB4), adenosine 5-triphosphate binding cassette subfamily B member 11 (ABCB11), retinal-binding protein (RALBP) or cytochrome P851 (CYP851) that are associated with resistance to mithramycin-induced hepatotoxicity.
* Patients must have had or refused first-line standard therapy for their malignancies.
* Patients must be 18 years or older with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, without evidence of unstable or decompensated myocardial disease. Patients must have adequate pulmonary reserve evidenced by forced expiratory volume 1 (FEV1) and diffusing capacity for carbon monoxide (DLCO) equal to or greater than 30% predicted; oxygen saturation greater than or equal to 92% on room air. Arterial Blood Gas (ABG) will be drawn if clinically indicated.
* Patients must have a platelet count greater than 100,000, an absolute neutrophil count (ANC) equal to or greater than 1500 without transfusion or cytokine support, a normal prothrombin time (PT)/partial thromboplastin time (PTT), and adequate hepatic function as evidenced by a total bilirubin of <1.5 times upper limits of normal (ULN) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 3 x ULN. Serum creatinine less than 3 or equal to 1.6 mg/ml, or creatinine clearance greater than 70 ml/min/1.73m^2.

Design:

* Simon Optimal Two Stage Design for Phase II Clinical Trials targeting an objective response rate (Response Evaluation Criteria in Solid Tumors (RECIST)) of 30%.
* Patients will be stratified based on location of primary disease (thoracic vs. extra-thoracic).
* Patients will receive 6 hour infusions of mithramycin at 30 -50 mcg/kg every day for 7 days, every 21 days (1 cycle). Three cycles will constitute one course of therapy. Those patients tolerating 30 mcg/kg infusions during the first cycle will receive subsequent cycles of mithramycin at a dose of 50 mcg/kg using the same infusion schedule.
* Following each course of therapy, patients will undergo restaging studies. Patients exhibiting objective response to therapy or stable disease by RECIST criteria will be offered an additional course of therapy.
* Patients exhibiting disease progression will be removed from study.
* Biopsies of index lesions will be obtained at baseline and on day 8 of the second cycle of therapy for analysis of molecular end-points.
* Pharmacokinetics will be assessed during cycle 1 and cycle 2 of the first course of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis: Patients with measurable inoperable, histologically confirmed primary lung and esophageal carcinomas, thymic neoplasms, germ cell tumors, malignant pleural mesotheliomas or chest wall sarcomas, as well as patients with gastric, colorectal or renal cancers and sarcomas metastatic to the thorax are eligible
* Histologic confirmation of disease in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), National Institutes of Health (NIH).
* Disease amenable to biopsy via percutaneous approach or other minimally invasive procedures such as thoracoscopy, bronchoscopy, laparoscopy, or gastrointestinal (GI) endoscopy
* Age >18
* Eastern Cooperative Oncology Group (ECOG) status 0-2.
* Patients must have had or refused first-line standard chemotherapy for their inoperable malignancies.
* Patients must have had no chemotherapy, biologic therapy, or radiation therapy for their malignancy for at least 30 days prior to treatment. Patients may have received localized radiation therapy to non-target lesions provided that the radiotherapy is completed 14 days prior to commencing therapy, and the patient has recovered from any toxicity. At least 3 half-lives must have elapsed since monoclonal antibody treatment. At least six weeks must have elapsed between mitomycin C or nitrosourea treatment.
* Patients must have adequate organ and marrow function as defined below:

  a) Hematologic and Coagulation Parameters:

  i. Peripheral absolute neutrophil count (ANC) greater than or equal to 1500/mm^3

ii. Platelets greater than or equal to 100,000/ mm^3 (transfusion independent)

iii. Hemoglobin greater than or equal to 8 g/dL (peripheral red blood count (PRBC) transfusions permitted)

iv. Prothrombin Time (PT)/Partial Thromboplastin Time (PTT) within normal limits (patient may be eligible for trial if abnormality is deemed clinically insignificant and cleared for protocol therapy by Hematology Consult Service)

b) Hepatic Function

i. Bilirubin (total) < 1.5 times upper limit of normal (ULN)

ii. Alanine aminotransferase (ALT) (Serum glutamic pyruvic transaminase (SGPT)) less than or equal to 3.0 times ULN

iii. Albumin > 2 g/dL

c) Renal Function

i. Creatinine within normal institutional limits or creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

ii. Normal ionized calcium, magnesium and phosphorus (can be on oral supplementation)

* Cardiac Function: Left ventricular ejection fraction (EF) >40% by Echocardiogram, multi-gated acquisition scan (MUGA), or cardiac magnetic resonance (MR).
* Ability of subject to understand, and be willing to sign informed consent.
* Female and male patients (and when relevant their partners) must be willing to practice birth control (including abstinence) during and for two months after treatment, if of childbearing potential during sexual contact with a female of childbearing potential.
* Patients must be willing to undergo 2 tumor biopsies

EXCLUSION CRITERIA:

* Patients with adenosine 5-triphosphate binding cassette subfamily B member 4 (ABCB4), adenosine 5-triphosphate binding cassette subfamily B member 11 (ABCB11), retinal-binding protein (RALBP) or cytochrome P851 (CYP851) genotypes associated with mithramycin-mediated hepatotoxicity.
* Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgment of the Principal Investigator (PI) would compromise the patients ability to tolerate protocol therapy or significantly increase the risk of complications
* Patients with cerebral metastases
* Patients with any of the following pulmonary function abnormalities will be excluded: forced expiratory volume (FEV), < 30% predicted; diffusing capacity for carbon monoxide (DLCO), < 30% predicted (post-bronchodilator); Oxygen saturation greater than 92% on room air. Arterial Blood Gas will be drawn if clinically indicated.
* Patients with evidence of active bleeding, intratumoral hemorrhage or history of bleeding diatheses, unless specifically occurring as an isolated incident during reversible chemotherapy induced thrombocytopenia
* Patients on therapeutic anticoagulation. Note: prophylactic anticoagulation (i.e. intraluminal heparin) for venous or arterial access devices is allowed
* Patients who are concurrently receiving or requiring any of the following agents, which may increase the risk for mithramycin related toxicities, such as hemorrhage:

  * Thrombolytic agents
  * Aspirin or salicylate-containing products, which may increase risk of hemorrhage
  * Dextran
  * Dipyridamole
  * Sulfinpyrazone
  * Valproic acid
  * Clopidogrel
* Lactating or pregnant females (due to risk to fetus or newborn, and lack of testing for excretion in breast milk)
* Patients with history of Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) due to potentially increased risk of mithramycin toxicity in this population
* Hypersensitivity to mithramycin
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Smoking-attributable mortality, years of potential life lost, and productivity losses--United States, 2000-2004. MMWR Morb Mortal Wkly Rep. 2008 Nov 14;57(45):1226-8. PMID 19008791
- [Background] Zhai R, Chen F, Liu G, Su L, Kulke MH, Asomaning K, Lin X, Heist RS, Nishioka NS, Sheu CC, Wain JC, Christiani DC. Interactions among genetic variants in apoptosis pathway genes, reflux symptoms, body mass index, and smoking indicate two distinct etiologic patterns of esophageal adenocarcinoma. J Clin Oncol. 2010 May 10;28(14):2445-51. doi: 10.1200/JCO.2009.26.2790. Epub 2010 Apr 12. PMID 20385987
- [Background] Wright CD, Kucharczuk JC, O'Brien SM, Grab JD, Allen MS; Society of Thoracic Surgeons General Thoracic Surgery Database. Predictors of major morbidity and mortality after esophagectomy for esophageal cancer: a Society of Thoracic Surgeons General Thoracic Surgery Database risk adjustment model. J Thorac Cardiovasc Surg. 2009 Mar;137(3):587-95; discussion 596. doi: 10.1016/j.jtcvs.2008.11.042. PMID 19258071

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 - 30 mcg/kg Thoracic Malignancy; Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy: Single agent intravenous (IV) mithramycin
  Mithramycin: 30 mcg/kg intravenous (IV) over 6 hours once daily for 7 days, to be repeated every 21 days (one cycle) until disease progression or unacceptable toxicity.
- Dose Level -1 - 25 mcg/kg Thoracic Malignancy; Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy: Single agent intravenous (IV) mithramycin
  Mithramycin: 25 mcg/kg intravenous (IV) over 6 hours once daily for 7 days, to be repeated every 21 days (one cycle).
Period: Overall Study
Arm/Group | Dose Level 1 - 30 mcg/kg Thoracic Malignancy | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy
Started | 2 | 2 | 10 | 2
Completed | 2 | 0 | 3 | 2
Not Completed | 0 | 2 | 7 | 0
Not completed — DLT, taken off therapy | 0 | 1 | 0 | 0
Not completed — Withdrew prior to treatment | 0 | 1 | 0 | 0
Not completed — Died on study | 0 | 0 | 2 | 0
Not completed — Did not complete 1 crse of therapy | 0 | 0 | 2 | 0
Not completed — Dose escalated | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was collected and is being reported for one participant that was enrolled in the 30 mcg/kg extra thoracic group but withdrew prior to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - 30 mcg/kg Thoracic Malignancy | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy | Total
Number analyzed (Participants) | 2 | 2 | 10 | 2 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 6 | 2 | 12
  >=65 years | 0 | 0 | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (1) | 34.5 (7.5) | 59.1 (9.65) | 50.5 (10.5) | 56.86 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 2 | 2 | 9 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 10 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 1 | 2 | 8 | 2 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 10 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Response (Complete Response + Partial Response)
Description: Objective response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesion, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 8 weeks until disease progression or unacceptable toxicity, over an average of 4 months.
Population: One participant in DL1 30 mcg thoracic died on study, one participant in DL1 30 mcg extra thoracic experienced a dose limiting toxicity and was taken off therapy, and 1 withdrew prior to trmt, two participants in DL1 25 mcg thoracic died on study, and two did not complete one course of therapy prior to treatment evaluation for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 30 mcg/kg Thoracic Malignancy | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy
Number analyzed (Participants) | 1 | 0 | 6 | 2
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 0 | 0 | 0 | 0
  Progressive Disease | 1 | 0 | 6 | 2

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approx. 9 mos & 6 days DL1 30 mcg/kg thoracic group, 2 mos & 16 days DL1 30 mcg/kg extra-thoracic group, 5 mos & 26 days DL-1 25 mcg/kg thoracic group, & 20 days DL-1 25 mcg/kg extra-thoracic group
Population: One participant was enrolled in the 30 mcg/kg extra thoracic group but withdrew prior to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 30 mcg/kg Thoracic Malignancy | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy
Number analyzed (Participants) | 2 | 1 | 10 | 2
Participants | 2 | 1 | 10 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 9 months and 6 days for the DL1 30 mcg/kg thoracic group, 2 months and 16 days for the DL1 30 mcg/kg extra-thoracic group, 5 months and 26 days for the DL-1 25 mcg/kg thoracic group, and 20 days for the DL-1 25 mcg/kg extra-thoracic group.
Description: One participant was enrolled in the 30 mcg/kg extra thoracic group but withdrew prior to treatment.
Arm/Group | Dose Level 1 - 30 mcg/kg Thoracic Malignancy | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Thoracic Malignancy | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1 | 2/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 2/10 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 10/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 30 mcg/kg Thoracic Malignancy (N=2) | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy (N=1) | Dose Level -1 - 25 mcg/kg Thoracic Malignancy (N=10) | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy (N=2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 30 mcg/kg Thoracic Malignancy (N=2) | Dose Level 1 - 30 mcg/kg Extra Thoracic Malignancy (N=1) | Dose Level -1 - 25 mcg/kg Thoracic Malignancy (N=10) | Dose Level -1 - 25 mcg/kg Extra Thoracic Malignancy (N=2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (2) | 9 (26) | 2 (5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 1 (1) | 9 (22) | 2 (5)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT01624090/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT01624090/ICF_001.pdf